CLINICAL TRIAL: NCT04951388
Title: A Phase II, Prospective, Double-blinded, Multi-Center Study to Evaluate the Safety, Tolerability, and Immunogenicity of the SARS CoV 2 Vaccine Candidate MVC COV1901 in Adolescents
Brief Title: A Study to Evaluate MVC-COV1901 Vaccine Against COVID-19 in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CT-COV-22
Record Dates: First submitted 2021-06-30; First posted 2021-07-06 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2021-08

CONDITIONS: Covid19 Vaccine
Keywords: Covid19 Vaccine
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVC-COV1901(S protein with adjuvant) (Experimental): S-2P protein with CpG and Aluminum Hydroxide/0.5mL
  Interventions: Biological: MVC-COV1901(S protein with adjuvant)
- MVC-COV1901(Saline) (Placebo Comparator): Saline/0.5 mL
  Interventions: Biological: MVC-COV1901(Saline)

INTERVENTIONS:
Biological: MVC-COV1901(S protein with adjuvant) — Approximately 330 participants will receive 2 doses of MVC-COV1901(S-2P protein with adjuvant) at Visit 2 (Day 1) and Visit 4 (Day 29) via intramuscular (IM) injection in the deltoid region
  Arms: MVC-COV1901(S protein with adjuvant)
Biological: MVC-COV1901(Saline) — Approximately 55 participants will receive 2 doses of MVC-COV1901(Saline) at Visit 2 (Day 1) and Visit 4 (Day 29) via IM injection in the deltoid region
  Arms: MVC-COV1901(Saline)

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of MVC-COV1901 vaccine compared to placebo in participants aged ≥ 12 to < 18 years.

DETAILED DESCRIPTION:
This is a Phase II, prospective, placebo-controlled, double-blinded (investigator/site staff and participants), multi-center study; the Sponsor will be blinded until the interim analysis. Participants aged ≥ 12 to < 18 years will be enrolled. All eligible participants will be randomized to receive either MVC-COV1901 or placebo in a 6:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant ≥ 12 to < 18 years of age at randomization.
* Body mass index (BMI) at or above the third percentile according to World Health Organization (WHO) BMI-for-age at the Screening Visit.
* Female participant must:

  1. Be either of non-childbearing potential, i.e. surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient);
  2. Or, if of childbearing potential, be abstinent or agree to use medically effective contraception from 14 days before screening to 30 days following the last injection of study intervention. Acceptable forms include:

  i. Implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system ii. Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
* Has a negative pregnancy test
* Participant is willing and able to comply with all required study visits and follow-up required by this protocol.
* Participant has not travelled overseas within 14 days of screening and will not have any oversea traveling throughout the study period.
* Participant and the participant's legal representative must understand the procedures of the study and provide written informed consent.

Exclusion Criteria:

* Pregnant or breast feeding or have plan to become pregnant in 30 days after last administration of study intervention.
* Currently receiving or received any investigational intervention within 30 days prior to the first dose of study intervention.
* Participant previously received a coronavirus vaccine.
* Administered any licensed live-attenuated vaccines within 28 days or other licensed non-live-attenuated vaccines within 7 days prior to the first dose of study intervention.
* Administered any blood product or intravenous immunoglobulin administration within 12 weeks prior to the first dose of study intervention.
* Currently receiving or anticipate to receive concomitant immunosuppressive or immune-modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg or equivalent) within 12 weeks prior to the first dose of study intervention.
* Currently receiving or anticipate to receive treatment with tumor necrosis factor (TNF)-α inhibitors, e.g. infliximab, adalimumab, etanercept within 12 weeks prior to the first dose of study intervention.
* Major surgery or any radiation therapy within 12 weeks prior to the first dose of study intervention
* Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ, bone marrow transplantation, or asplenia.
* Personal or family (linear or collateral relatives by blood within two generations) history of Guillain-Barré syndrome.
* A history of malignancy with potential risk for recurrence after curative treatment, or current diagnosis of or treatment for cancer (exceptions are squamous and basal cell carcinomas of the skin and treated uterine cervical carcinoma in situ, at the discretion of the investigator).
* Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
* Participant with ongoing acute diseases or serious medical conditions which will interfere with adherence to study requirements, or the evaluation of any study endpoint. Acute diseases or serious medical conditions include cardiovascular, pulmonary, hepatic, neurologic, metabolic, renal, psychiatric condition (e.g. alcoholism, drug abuse, anorexia or severe depression), current severe infections, autoimmune disease, medical history, physical findings, or laboratory abnormality that in the investigators' opinion are not in stable condition and participating in the study could adversely affect the safety of the participant.
* Participant with previous known SARS-CoV-1 or 2 infection.
* Participant with a history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the MVC-COV1901.
* Body (oral, rectal, or ear) temperature ≥ 38.0°C or acute illness (not including minor illnesses such as diarrhea or mild upper respiratory tract infection at the discretion of the investigator) within 2 days before the first dose of study intervention.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 399 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events(AEs) [Safety and Tolerability] | Day 1 to 28 days after the second vaccination
  To evaluate the incidence of Adverse Events(AEs) of MVC-COV1901 from Visit 2 (Day 1) to Visit 6 (28 days after the second dose of study intervention) in terms of the number and percentage of participants with the occurrence of:
  Solicited local AEs (up to 7 days after each dose of study intervention) Solicited systemic AEs (up to 7 days after each dose of study intervention) Unsolicited AEs (up to 28 days after each dose of study intervention) AE of Special Interest (AESI) Vaccine-Associated Enhanced Disease(VAED) Serious adverse events (SAEs)
Immunogenicity of MVC-COV1901-1 | Day 1 to 28 days after the second vaccination
  To evaluate the immunogenicity of MVC-COV1901, as compared to placebo, in terms of neutralizing antibody titers.
  The neutralizing antibody titers at Visit 6 (28 days after the second dose of study intervention) in terms of:
  -Geometric mean titers (GMT)
Immunogenicity of MVC-COV1901-2 | Day 1 to 28 days after the second vaccination
  To evaluate the immunogenicity of MVC-COV1901, as compared to placebo, in terms of neutralizing antibody titers.
  The neutralizing antibody titers at Visit 6 (28 days after the second dose of study intervention) in terms of:
  -Seroconversion rate (SCR)
Immunogenicity of MVC-COV1901-3 | Day 1 to 28 days after the second vaccination
  To evaluate the immunogenicity of MVC-COV1901, as compared to placebo, in terms of neutralizing antibody titers.
  The neutralizing antibody titers at Visit 6 (28 days after the second dose of study intervention) in terms of:
  -GMT ratio

SECONDARY OUTCOMES:
Incidence of Adverse Events(AEs) [Safety and Tolerability] | Day 1 to 180 days after the second vaccination
  To evaluate the Incidence of Adverse Events(AEs) of MVC-COV1901 over the study period in terms of the number and percentage of participants with the occurrence of:
  >= Grade 3 AE AE of Special Interest (AESI) Vaccine-Associated Enhanced Disease(VAED) Serious adverse events (SAEs)
Immunogenicity of MVC-COV1901-1 | Day 1 to 180 days after the second vaccination
  To evaluate the immunogenicity of MVC-COV1901, as compared to placebo, in terms of antigen-specific immunoglobulin titers and neutralizing antibody titers.
  The antigen-specific immunoglobulin titers and neutralizing antibody titers at Visit 4 (28 days after the first dose of study intervention), Visit 6 (28 days after the second dose of study intervention), Visit 8 (90 days after the second dose of study intervention) and Visit 9 (180 days after the second dose of study intervention) in terms of:
  -GMT
Immunogenicity of MVC-COV1901-2 | Day 1 to 180 days after the second vaccination
  To evaluate the immunogenicity of MVC-COV1901, as compared to placebo, in terms of antigen-specific immunoglobulin titers and neutralizing antibody titers.
  The antigen-specific immunoglobulin titers and neutralizing antibody titers at Visit 4 (28 days after the first dose of study intervention), Visit 6 (28 days after the second dose of study intervention), Visit 8 (90 days after the second dose of study intervention) and Visit 9 (180 days after the second dose of study intervention) in terms of:
  -SCR
Immunogenicity of MVC-COV1901-3 | Day 1 to 180 days after the second vaccination
  To evaluate the immunogenicity of MVC-COV1901, as compared to placebo, in terms of antigen-specific immunoglobulin titers and neutralizing antibody titers.
  The antigen-specific immunoglobulin titers and neutralizing antibody titers at Visit 4 (28 days after the first dose of study intervention), Visit 6 (28 days after the second dose of study intervention), Visit 8 (90 days after the second dose of study intervention) and Visit 9 (180 days after the second dose of study intervention) in terms of:
  -GMT ratio

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Huang, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (5):
- Taiwan (5):
  - Mackay Memorial Hospital Hsinchu, Hsinchu
  - Chang-Guang Memorial Hospital Lin-Kou, Taipei
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hospital-HsinChu, Taipei
  - National Taiwan University Hosptial, Taipei

REFERENCES:
- [Derived] Liu LT, Chiu CH, Chiu NC, Tan BF, Lin CY, Cheng HY, Lin MY, Lien CE, Chen C, Huang LM. Safety and immunogenicity of SARS-CoV-2 vaccine MVC-COV1901 in Taiwanese adolescents: a randomized phase 2 trial. NPJ Vaccines. 2022 Dec 16;7(1):165. doi: 10.1038/s41541-022-00589-4. PMID 36526640